CLINICAL TRIAL: NCT05679713
Title: Next-generation, Integrative, and Personalized Risk Assessment to Prevent Recurrent Heart Failure Events: the ORACLE Study
Acronym: ORACLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Josep Comín, Prof. Josep Comín-Colet, MD, PhD, Hospital Universitari de Bellvitge
Other Study IDs: PI21/00264
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
Keywords: Machine Learning; Multi-Omics Approaches; Outcomes Research; Patient-Centered Information
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comprehensive risk assessment algorithm — Risk assessment algorithm including clinical and patient-centered information and a novel RNA-based biomarkers using next-generation sequencing technology.

SUMMARY:
The aim of this study is to develop and validate an improved, comprehensive risk assessment algorithm integrating blood RNA-based biomarkers, clinical, and patient-centered data and to assess the incremental predictive value (discrimination and reclassification) compared to a traditional risk model (change in the c-statistics for prediction of the primary endpoint).

DETAILED DESCRIPTION:
The ORACLE study is a multicenter, observational, prospective, cross-sectional and longitudinal study integrated by 3 different cohorts for 1) RNA biomarker discovery (60 nested case-control sample), 2) model derivation (516 nested case-control sample) and 3) external validation (new prospective cohort of 558 consecutive patients recruited in 4 hospital centers) according to a TRIPOD Statement type 3 analysis. In total 1134 consecutive patients with a HF hospitalization or urgent HF visit < 30 days before inclusion and followed for 6 months will be studied.

This study include the discovery of novel RNA-based biomarkers using next-generation sequencing technology to define and validate a new biomarker set and clinical and patient-centered risk determinants definition. A new model will be constructed; training and internal validation in the derivation cohort using machine learning methods, and finally an external validation of the new next generation integrative risk assessment model will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients with a recent (<30 days) acute decompensation of HF requiring intravenous diuretic therapy (either hospitalized or in ambulatory care) or intensification of oral diuretics (ambulatory care).
* HF diagnosis according to European Society of Cardiology (ESC) criteria.
* Written informed consent
* Patients receiving oral standard medication for chronic HF.

Exclusion Criteria:

* Age<18 years old.
* Death before hospital discharge.
* The patient is unable or unwilling to give the informed consent to participate.
* Unstable patients with signs of fluid overload or low cardiac output at the moment of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The external validation cohort will be a multicenter, observational, prospective, cross-sectional and longitudinal cohort recruited for the specific purpose of the ORACLE study. The investigators plan to recruit patients with a recent (<30 days) acute HF event and follow them for 180 days. The study will be conducted in 4 different hospitals (University Hospital Bellvitge, Viladecans General Hospital, Vic General Hospital and Igualada General Hospital) covering a total healthcare area of > 650.000 inhabitants.
Sampling Method: Non-Probability Sample
Enrollment: 1134 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the model performance of the comprehensive risk assessment algorithm with a traditional risk model to predict HF related hospitalizations or all-cause death | 6 months
  To compare in an external validation cohort of patients a recent acute HF event, the performance (discrimination, additive predictive value, and reclassification ability) of a comprehensive risk assessment algorithm with the performance of a traditional risk model to predict the occurrence of the primary composite clinical end-point of HF related hospitalizations (readmissions) or all-cause death at 180 days after hospital discharge or after an urgent HF visit (acute HF event requiring intravenous administration of diuretics without admission).

SECONDARY OUTCOMES:
To compare the model performance of the comprehensive risk assessment algorithm with a traditional risk model to predict the occurrence of HF-related hospitalizations (readmissions) or all-cause death at 30, and 90 days after hospital discharge. | 6 months
  The admission will be considered as HF-related if it suits with one of the following conditions:
  * Cardiovascular cause hospitalization
  * Complication directly related with prior HF admission
  * Decompensation of prior disease or comorbidity
To compare the model performance of the comprehensive risk assessment algorithm with a traditional risk model to predict the occurrence of HF-related hospitalizations (readmissions) at 30, 90, and 180 days after hospital discharge. | 6 months
To compare the model performance of the comprehensive risk assessment algorithm with a traditional risk model to predict the occurrence of all-cause death at 30, 90, and 180 days, after hospital discharge. | 6 months

OTHER OUTCOMES:
Explore the performance (sensibility and specificity) of the developed model according gender, LVEF (preserved or reduced left ventricle ejection fraction), comorbidity burden (Charlson Comorbidity Index) and frailty. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No